CLINICAL TRIAL: NCT04983160
Title: Crossover Clinical Trial, Randomized, Double Blind, Placebo Controlled Trial. Modulation of Cellular Mediators and Repair Endothelial Damage in Patients With Chronic Renal Disease Through Inhibition of Xanthine Oxidase
Brief Title: Crossover Clinical Trial, Randomized, Double Blind, Placebo Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PI12/01866
Record Dates: First submitted 2015-03-31; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2015-03

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; allopurinol; CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allopurinol (Active Comparator)
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol — Allopurinol
  Arms: Allopurinol
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of inhibiting xanthine oxidase with allopurinol in patients with chronic kidney disease in asymptomatic hyperuricemia endothelial injury and vascular repair mechanisms.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effect of inhibiting xanthine oxidase with allopurinol in patients with chronic kidney disease in asymptomatic hyperuricemia endothelial injury and vascular repair mechanisms, evaluating the plasma concentration of angiogenic factors, microparticles of endothelial cells and the cell number circulating endothelial progenitor.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing and able to give informed consent for participation in the study
* Ability to understand study procedures and to comply with it for the duration of the study.
* Subjects of both sexes, the age range between 18 and 70 years old.
* Serum uric acid above 7 mg / dl.
* Estimated glomerular filtration rate by MDRD abbreviated formula less than 60 ml / min / 1.73 m2 and above 15 ml / min / 1.73 m2.
* Stability of renal function (serum creatinine increase without exceeding 50% in the three months before the start of the study).
* Clinically stable in terms of no hospitalizations of cardiovascular events in the 3 months before the study began.

Exclusion Criteria:

* Drop active in the 60 days prior to study initiation.
* Use of allopurinol within 60 days preceding baseline
* Active infections within 30 days prior to baseline.
* Patients with systemic inflammatory disease
* Infection with HIV, Hepatitis C and Hepatitis B.
* History of cancer within 5 years prior to the first dose of study medication
* Chronic liver disease.
* Immunosuppressive therapy.
* Pregnant women, breastfeeding or planning to become pregnant.
* Allergy or sensitive to allopurinol.
* Addiction to drugs or alcohol, in the opinion of the investigator, may interfere with compliance with study requirements.
* Inability or unwillingness of the individual or legal guardian or representative to give written informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-02-26 (Actual); Primary Completion 2016-04-29 (Actual); Study Completion 2016-04-29 (Actual)

PRIMARY OUTCOMES:
Circulating endothelial progenitor cells concentration and microparticles derived from endothelial cells | Data collected after 4 weeks, 8 weeks and 12 weeks.
  Effect of inhibiting xanthine oxidase with allopurinol in patients with CKD

SECONDARY OUTCOMES:
Level of oxidative stress | After patient visit (0 weeks, 4, 8 and 12 weeks)
  Evaluated through quantification of oxygen-reactive species
Level of micro inflammation | After patient visit (0 weeks, 4, 8 and 12 weeks)
  Evaluated through quantification of C-reactive protein, proinflammatory cytokines, CD14+ and CD16+ monocytes
Level of endothelial dysfunction | After patient visit (0 weeks, 4, 8 and 12 weeks)
  Endothelium-dependant vasodilation in response to ischemia evaluated through changes in capillar flux using Doppler laser PeriFlux system 5000
Blood pressure | Each visit (0 weeks, 4 weeks, 8 weeks and 12 weeks) for 24 hours
Glomerular filtration ratio | After patient visit (0 weeks, 4 weeks, 8 weeks and 12 weeks)
  Estimated through MDRD-4 y Cockroft-Gault.
Microalbuminuria / Proteinuria | Daily, using first urine of the day as a sample.
  Evaluated through albumin/creatinin ratio and protein/creatinine ratio

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Santamaría, MD, Principal Investigator — Hospital Universitario Reina Sofía
Locations (1):
- Hospital Universitario Reina Sofía de Córdoba, Córdoba, Spain